CLINICAL TRIAL: NCT06570512
Title: Evaluation of the Transcutaneous Electrical Nerve Stimulation of the Posterior Tibial Nerve in the Treatment of Premature Ejaculation: A Randomized Controlled Trial
Brief Title: Transcutaneous Electrical Nerve Stimulation for the Treatment of Premature Ejaculation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Department of Andrology & STDs Kasr AlAiny Cairo University (Unknown)
Responsible Party: Principal Investigator, Mahmoud Fawzy Ghaly, Doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TPTNS for PE
Record Dates: First submitted 2024-08-01; First posted 2024-08-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Transcutaneous Electrical Nerve Stimulation; Premature Ejaculation
Keywords: premature ejaculation; transcutaneous electrical nerve stimulation; posterior tibial nerve
MeSH Terms: conditions — Premature Ejaculation | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- transcutaneous posterior tibial nerve stimulation (TPTNS) (Experimental): TPTNS group underwent ten sessions of electrical stimulation along the course of the posterior tibial nerve behind the medial malleoli using cup electrodes, with a width pulse of 250 microseconds, and a frequency of 20 Hz
  Interventions: Device: transcutaneous posterior tibial nerve stimulation
- sham transcutaneous electrical nerve stimulation (TENS). (Active Comparator): TENS group used a sham device with the same parameters, but the electrodes were placed behind the lateral malleoli with underpowered amplitudes.
  Interventions: Device: transcutaneous posterior tibial nerve stimulation

INTERVENTIONS:
Device: transcutaneous posterior tibial nerve stimulation — Over three weeks, the TPTNS group underwent ten sessions of electrical stimulation along the course of the posterior tibial nerve behind the medial malleoli using cup electrodes, with a width pulse of 250 microseconds, and a frequency of 20 Hz. The TENS group used a sham device with the same parameters, but the electrodes were placed behind the lateral malleoli with underpowered amplitudes.
  Other Names: sham transcutaneous electrical nerve stimulation (TENS).

SUMMARY:
Premature ejaculation (PE) is the most prevalent male sexual dysfunction. The currently approved treatments are intolerable to patients due to their side effects.

the investigatorsconducted a blinded randomized controlled trial to evaluate the efficacy and safety of transcutaneous posterior tibial nerve stimulation (TPTNS) for the treatment of PE.

5o male patients complaining of PE with intravaginal ejaculation latency time (IELT) of less than 2 minutes were randomized into two equal groups to receive either TPTNS or sham transcutaneous electrical nerve stimulation (TENS). TPTNS group underwent ten sessions of electrical stimulation of the posterior tibial nerve using a frequency of 20 Hz and a pulse width of 250 microseconds. The primary outcomes were IELT which was calculated by the patient's digital hand watch, and the Arabic index of premature ejaculation (AIPE).

DETAILED DESCRIPTION:
Trial design A single blinded randomized controlled trial was used, and the ratio of allocation was 1:1.

Between 2022 and 2023, this study was conducted on (50) male patients attending the outpatient clinic of Andrology, Kasr Al Ainy Hospital, Cairo University to evaluate the efficacy and safety of transcutaneous posterior tibial nerve stimulation (TPTNS) to delay ejaculation in PE patients compared to sham transcutaneous electrical nerve stimulation (TENS).

Patients The participants included in this study were married males with stable and continuous marital relationships, diagnosed with premature ejaculation based on the International Society for Sexual Medicine (ISSM-International Society for Sexual Medicine) : (a) within the 1-2 minutes after penetration, the ejaculation always or almost always starts; (b)in all or almost all penetrations, the patient cannot delay the ejaculation; (c) PE generate negative consequences on the patients, such as discomfort, frustration, stress, and/or sexual intimacy avoidance, and the patient did not take the treatment for PE in the previous 14 days. Patients were excluded if they had erectile dysfunction (measured by the International Index of Erectile function-ILEF-5 questionnaire), inhibited male orgasm, reduced sexual desire, uncontrolled physical illness, active genitourinary tract infection (confirmed by two glasses of urine according to Modified Meares-Stamey technique), mental disorders affecting ejaculatory function such as anxiety, depression, and schizophrenia, history of alcohol or drug abuse. To exclude chronic prostatitis patients, the expressed prostatic secretions after prostatic massage were subjected to microscopic examination. Before conducting the study, informed consent was obtained from each patient.

The applied technique Over three weeks, the TPTNS group underwent ten sessions of electrical stimulation along the course of the posterior tibial nerve behind the medial malleoli using cup electrodes, with a width pulse of 250 microseconds, and a frequency of 20 Hz. The TENS group used a sham device with the same parameters, but the electrodes were placed behind the lateral malleoli with underpowered amplitudes.

Outcome measures Before and after treatment, the patients were asked to answer the Arabic Index of premature ejaculation questionnaire (AIPE) which evaluates seven items: time to ejaculation, hard erections for sufficient intercourse, control, sexual desire, satisfaction for the patient and partner, anxiety, or depression. Also, the intravaginal ejaculation latency time (IELT) was calculated using the digital hand watch, as the patients were instructed to count the time between intromission and ejaculation, and to repeat this procedure in one to two coital occasions per week over three weeks after receiving either TPTNS or TENS. The ISSM defined an IELT threshold of 2 minutes as the cut-off point for PE. The treatment success was defined as a decrease in PE severity and an improvement in AIPE score.

ELIGIBILITY:
Inclusion Criteria:

* married males
* with stable and continuous marital relationships
* diagnosed with premature ejaculation based on the International Society for Sexual Medicine (ISSM-International Society for Sexual Medicine) : (a) within the 1-2 minutes after penetration, the ejaculation always or almost always starts; (b)in all or almost all penetrations, the patient cannot delay the ejaculation; (c) PE generate negative consequences on the patients, such as discomfort, frustration, stress, and/or sexual intimacy avoidance
* and the patient did not take the treatment for PE in the previous 14 days

Exclusion Criteria:

* Patients were excluded if they had erectile dysfunction (measured by the International Index of Erectile function-ILEF-5 questionnaire),
* inhibited male orgasm
* reduced sexual desire
* uncontrolled physical illness
* active genitourinary tract infection (confirmed by two glasses of urine according to Modified Meares-Stamey technique)
* mental disorders affecting ejaculatory function such as anxiety, depression, and schizophrenia, history of alcohol or drug abuse

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-12-09 (Actual)

PRIMARY OUTCOMES:
Intravaginal ejaculation latency time (ILET) | at the baseline (before starting the treatment sessions), then at 3 weeks (by the end of treatment) and finally 2 months later for follow up
  was calculated using the digital hand watch. The patients were instructed to count the time between intromission and ejaculation, and to repeat this procedure in one to two coital occasions per week over three weeks of receiving sessions and to continue for 2 months after end of sessions.
Score of Arabic index of premature ejaculation (AIPE) | at the baseline (before starting the treatment sessions), then at 3 weeks (by the end of treatment) and finally 2 months later for follow up
  Seven item questionnaire developed by Arafa & Shamloul in 2007 that evaluates sexual desire, hard erections for sufficient intercourse, time to ejaculation, control, satisfaction for the patient and partner, anxiety or depression.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Cairo University, Cairo, Giza Governorate
  - Faculty Of Medicine, Cairo University, Cairo

IPD SHARING:
Plan to Share IPD: Undecided